CLINICAL TRIAL: NCT04416022
Title: Cervical Gland Area as a Predictor of Success of Labour Induction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, SAAR AHARONI MD, Dr. Saar Aharoni, Rambam Health Care Campus
Other Study IDs: 0711-19-RMB
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Induced Vaginal Delivery
Keywords: Labour induction; Cervical glandular area

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound examination — Women that are planned for labour induction, will undergo a routine ultrasound examination prior to the initiation of the induction process.

SUMMARY:
Women who fulfil the inclusion criteria and who are planned for labour induction will be recruited. Bishop score, cervical length, and the presence of cervical glandular area (CGA) will be documented for every patient up to 12 hours prior to the induction process, and patient information and maternal and neonatal outcome will be documented following the delivery.

DETAILED DESCRIPTION:
Patient consent to participate in the study will be retrieved following the medical decision of labor induction and the mode of induction and following the patient consent to the induction.

Bishop score, cervical length, and the presence of cervical glandular area (CGA) will be documented for every patient up to 12 hours prior to the induction process.

The method of induction, data regarding patient demographics, the progress of labor, and the maternal and neonatal outcome will be documented following the delivery.

ELIGIBILITY:
Inclusion Criteria:

* Singleton and twins' pregnancies
* Pregnancy 34-41 weeks of gestation
* Vertex presentation
* Induction methods (Oxytocin, prostaglandin 1 (PGE1), prostaglandin 2 (PGE2), double balloon catheter, rupture of memebrane (ROM)

Exclusion Criteria:

* Intrauterine fetal demise (IUFD)
* Contraindication to vaginal delivery
* Status post cervical cerclage
* Previous attempt of labor induction
* History of cervical surgery
* Active vaginal bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who are planned form labour induction
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-07 (Estimated); Primary Completion 2022-06-07 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
Onset of active labour | Up to delivery
  Percent of patients that reached the active stage of labour (defined as measurement of cervical dilation of greater than 6 cm)

SECONDARY OUTCOMES:
Time from Induction to second stage | Up to delivery
  Duration of time from initiation of labpur induction to cervical dilation of 10cm
Time from Induction to delivery | Up to delivery
  Duration of time from initiation of labpur induction to delivery
Rate of vaginal delivery | Up to delivery
  The rate of patient that deliver vaginally including instrumental deliverires
Neonatal outcome - PH | Up to 10 minutes from delivery
  The fetal arterial pH measuerment following the delivery
Neonatal outcome - APGAR (Apearance, Pulse, Grimace, Activity, Respiration score) | Up to 5 minutes from delivery
  The fetal APGAR score as recieved by pediatrician
Neonatal outcome - NICU (Neonatal Intensive Care Unit) admission | Up to 48 hours from delivery
  Percent of neonated that requiered NICU admission

IPD SHARING:
Plan to Share IPD: Undecided